CLINICAL TRIAL: NCT05657171
Title: "Effect of Cyproterone Acetate / Ethinyl Estradiol Combination on Periodontal Tissue and High Sensitivity C- Reactive Protein Levels in Women With Polycystic Ovary Syndrome Having Gingivitis."
Brief Title: "Effect of CPA/EE Drug on Periodontal Tissue and hsCRP Levels in PCOS Patients With Gingivitis
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Dr Ridhima perio/22/25
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Cyproterone Acetate; Cyproterone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCOS +GINGIVITIS: FEMALE PATIENTS WITH PCOS AND GINGIVITIS ON CPA/EE DRUG REGIMEN
  Interventions: Drug: cyproterone Acetate/Ethinyl Estradiol Combination

INTERVENTIONS:
Drug: cyproterone Acetate/Ethinyl Estradiol Combination — cyproterone acetate (CPA) 2 mg, combined with EE 35 µg.
  Other Names: Diane 35

SUMMARY:
PCOS is a widely reported condition among young female population and anti-androgen agents are increasingly being used as part of the medical management of such cases. However, Clinical studies have reported higher prevalence of gingival inflammation, loss of attachment and gingival enlargement in women taking hormone based oral contraceptives. Additionally, CPA has been reported to have an osteoclastic action. Therefore, it is necessary to explore the effects of these medications on the periodontal condition of PCOS patients having gingivitis, who already are pre-disposed to systemic inflammation. Therefore, the present study aims to longitudinally evaluate the effect of CPA/EE combination regimen on the periodontal status of female patients diagnosed with PCOS with pre-existing gingivitis..

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a complex endocrine, reproductive and metabolic condition, affecting women of reproductive age globally with a worldwide prevalence ranging from 5-15%. PCOS is associated with low-grade systemic inflammation and is characterised by elevation of multiple markers of inflammation such as C-reactive protein (CRP), proinflammatory cytokines and chemokines, white blood cell count as well as increased oxidative stress.CRP is a serologic marker of systemic inflammation that has been associated with increased risk for various systemic diseases. Gingivitis has been linked to elevated CRP levels. Also, elevated C-reactive protein (CRP) levels are associated with PCOS.

It has been hypothesised that PCOS might exacerbate the periodontal condition that is caused by dental plaque, through various pathophysiological links, namely, low-grade systemic inflammation, oxidative stress, insulin resistance (IR), advanced glycation end products (AGE), and systemic hormonal levels. Evidence has suggested that periodontal disease causes chronic subclinical inflammation leading to Insulin resistance, initiating the development of type 2 diabetes, which in turn is a prominent feature in PCOS. Hence, a two-way relationship between PCOS and periodontal disease is currently being explored.

The imbalance of Luteinizing Hormone(LH) and Follicle Stimulating Hormone (FSH) in women with PCOS explains the rationale for treatment with combined hormonal treatment.One such therapy is cyproterone acetate (CPA) 2 mg, combined with EE 35 µg. CPA is a steroidal antiandrogen progestogen while EE is one of the most potent oral estrogens .EE enhances the action of CPA by increasing sex hormone binding globulin (SHBG) levels, which leads to a reduction in free testosterone and thus adds to the antiandrogenic action of CPA.

Receptors for estrogen have been demonstrated in the gingiva and periodontal connective tissue cells .The use of hormonal contraceptives by women has been reported to influence periodontal disease progression. While the effects of different contraceptive combinations and/or oral hypoglycemics on the periodontal condition of female patients diagnosed with PCOS has been explored, the specific drug combination of CPA/EE has not been studied in detail as yet. Therefore, the present study aims to longitudinally evaluate the effect of CPA/EE combination regimen on the periodontal status of female patients diagnosed with PCOS with pre-existing gingivitis.

The present cohort study is conducted in the Department of periodontology, Post Graduate Institute of Dental Sciences, Rohtak in collaboration with Department of Obstetrics and Gynaecology Post Graduate Institute of Medical Sciences, Rohtak over a period of 12-14 months. The study population comprised of female patients diagnosed with PCOS having gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Females of age group (15-40yrs) diagnosed with PCOS. The diagnosis of PCOS will be according to Rotterdam criteria, when any two out of the following three abnormalities will be present:

  1. clinical (hirsutism, acne or acanthosis nigricans) and/or biochemical (raised testosterone) hyperandrogenism ;
  2. chronic anovulation (oligomenorrhoea or amenorrhea); and
  3. polycystic ovaries on ultrasound (one or both ovaries demonstrate 12 or more follicles measuring 2 to 9 mm in diameter or the ovarian volume exceeds 10 cubic cm on pelvic ultrasound) from department of Obstetrics and Gynaecology, Post Graduate Institute of Medical Sciences, Rohtak.
* presence of ≥20 natural teeth
* BMI (18.5 - 24.9)
* Presence of gingivitis

  1. Gingivitis with intact periodontium - BOP ≥ 10% of sites , with pockets ≤ 3mm, no probing attachment loss and no radiographic bone loss .
  2. Gingivitis with reduced periodontium - BOP ≥ 10% of sites , with pockets ≤ 3mm with possible probing attachment loss and possible radiographic bone loss.
  3. Localized gingivitis - 10 to 30%of bleeding sites.
  4. Generaized gingivitis - more than 30% of beeding sites.

Exclusion Criteria:

* Previous history of androgen-secreting tumors, congenital adrenal hyperplasia , hyperprolactinemia, or any thyroid dysfunction
* Patients with chronic inflammatory disease such as nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, or active cancer within the past 5 years
* Smokers and alcoholics,
* History of systemic antibiotics or oral contraceptives usage within last 3 months,
* Periapical pathology or other oral inflammatory conditions and any periodontal treatment within 6 months prior to study

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Female patients diagnosed with PCOS having gingivitis
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 6 months
  BOP will be recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing
CLINICAL ATTACHMENT LEVEL (CAL) | 6 months
  Clinical Attachment Level will be measured as the distance between the base of the clinical pocket and the cemento-enamel junction(CEJ).Measurements will be made at 6 sites of involved tooth- mesio-buccal, mid- buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual using UNC-15 probe. Measurements will be rounded to the nearest whole millimetre. Distance of base of the pocket from gingival margin, distance of free gingival margin from CEJ.
PROBING POCKET DEPTH (PPD) | 6 months
  Probing pocket depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of involved tooth - mesio-buccal, mid-buccal, disto-buccal, mesio- lingual, mid-lingual, disto-lingual. Measurements will be rounded to the nearest whole millimetre.
hsCRP Levels | 6 months
  Blood samples for the investigation of serum hsCRP will be collected after overnight fasting. Venous blood from the antecubital vein will be collected after applying a tourniquet in plain tubes without additive. Serum hsCRP levels will be assessed using a kit‡ with high sensitivity methodology in an auto-analyzer§ according to the manufacturer's instructions. The test principle will be particle-enhanced immune- turbidimetric assay, in which human CRP agglutinates with latex particles coated with monoclonal anti-CRP antibodies.

SECONDARY OUTCOMES:
Plaque index | 6 months
  Plaque index by Silness and Loe (1964) will be used for assessment of plaque. For the scoring, a mouth mirror, an explorer and a light source will be used on air dried teeth and gingiva.
Gingival index | 6 months
  Gingival Index by Loe and Silness (1963) will be used for assessment of severity of gingival inflammation. For the scoring, a mouth mirror, a probe and a light source will be used on air dried teeth and gingiva.
Gingival recession | 6 months
  Gingival recession is defined as the apical shift of the gingival margin with respect to the cemento-enamel junction (CEJ); it is associated with attachment loss and with exposure of the root surface to the oral environment

CONTACTS AND LOCATIONS:
Overall Officials: Ridhima Singhal, BDS, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No